CLINICAL TRIAL: NCT06991348
Title: Multicenter, Active-controlled, Randomized, Double-blind, Clinical Trial for the Comparative Evaluation of Acid Suppression and Symptom Management of Gastroesophageal Reflux Disease With the Administration of Tegoprazan or Pantoprazole: TOP-GERD
Brief Title: Clinical Trial for the Comparative Evaluation of Acid Suppression and Symptom Management of Gastroesophageal Reflux Disease With the Administration of Tegoprazan or Pantoprazole
Acronym: TOP-GERD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Carnot Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRN-GA-01-2022
Record Dates: First submitted 2025-05-20; First posted 2025-05-27 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; pantoprazole; tegoprazan; P-CAB; PPI
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — tegoprazan; Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-erosive GERD - Test product (Experimental): Non-erosive GERD - Tegoprazan
  Interventions: Drug: Tegoprazan
- Non-erosive GERD - Comparator (Active Comparator): Non-erosive GERD - Pantoprazole
  Interventions: Drug: Pantoprazole
- Erosive GERD - Test product (Experimental): Erosive GERD - Tegoprazan
  Interventions: Drug: Tegoprazan
- Erosive GERD - Comparator (Active Comparator): Erosive GERD - Pantoprazol
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Tegoprazan — Tegoprazan 50 mg daily for 28 days
  Arms: Erosive GERD - Test product; Non-erosive GERD - Test product
Drug: Pantoprazole — Pantoprazole 40 mg daily for 28 days
  Arms: Erosive GERD - Comparator; Non-erosive GERD - Comparator

SUMMARY:
The objective of this clinical trial is to compare which of the two drugs best resolves symptoms in patients diagnosed with erosive and non-erosive gastroesophageal reflux disease, adult males and females. The main question is What is the proportion of patients with resolution of the main symptoms of gastroesophageal reflux disease at four weeks of treatment with pantoprazole vs tegoprazan.

ELIGIBILITY:
Inclusion Criteria:

* With endoscopic diagnosis of GERD or NERD (endoscopy ≤ 15 days old)
* With positive impedance pHmetry results (pHmetry ≤ 15 days old)
* With recurrent symptoms of heartburn and regurgitation for a previous period ≥ 3 months old

Exclusion Criteria:

* With known hypersensitivity to tegoprazan, pantoprazole, or any of the components of each formulation
* Subjects with concomitant administration of atazanavir, nelfinavir or rilpivirine
* Nephropathic and/or hepatopathic subjects (including non-alcoholic hepatitis)
* Subjects with upper gastrointestinal tract bleeding
* Subjects with gastric and/or duodenal ulcer 2 months prior to screening
* Subjects with a history of esophageal or gastric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with resolution of the main symptoms of gastroesophageal reflux disease | From enrollment to the end of treatment at 4 weeks
  Carlsson-Dent Questionnaire. These tool consists of 7 multiple-choice questions, using a cut-off point ≥ 4 to be considered positive, which qualitatively assesses symptoms associated with GERD and triggering factors such as diet, posture and medications used.

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Remes-Troche, Dr, Principal Investigator — Digestive Physiology and Motility Lab, Instituto de Investigaciones Médico Biológicas, Veracruz , México
Locations (2):
- Mexico (2):
  - Gastrologen S.A. de C.V., Mexico City, Mexico City
  - Saluz Investigación, S.C., Boca del Río, Veracruz

IPD SHARING:
Plan to Share IPD: No
Only IPD used in the results publication

REFERENCES:
- [Background] Cho YK, Kim JH, Kim HS, Kim TO, Oh JH, Choi SC, Moon JS, Lee SK, Jung SW, Kim SS, Jung HK, Lee SP, Cheon GJ, Park MI, Jung HY, Ko KH, Sung IK, Lee SH, Lee JY, Lee ST, Rhee PL, Kim N, Hong SJ, Kim HJ, Kim GH, Lee KJ, Kim SK, Shin WG, Lee OY. Randomised clinical trial: comparison of tegoprazan and lansoprazole as maintenance therapy for healed mild erosive oesophagitis. Aliment Pharmacol Ther. 2023 Jan;57(1):72-80. doi: 10.1111/apt.17255. Epub 2022 Oct 31. PMID 36314172